CLINICAL TRIAL: NCT06123572
Title: A Randomized, Double Blind, Two Arm, Parallel, Placebo-Controlled, Safety and Efficacy Study of Anti-Ageing and Skin Brightening Gel
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Anti-Ageing and Skin Brightening Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Green Mountain Biotech Limited (Unknown)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator-Medical Director, NovoBliss Research Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB230027-GB
Record Dates: First submitted 2023-10-26; First posted 2023-11-09 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Wrinkle; Pigment Skin; Aging
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Intervention Model Description: This is a Randomized, Interventional, Prospective, Double Blind, Two Arm, Comparative, Parallel, Placebo-Controlled, Safety and Efficacy Study
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomly assigned in as 1:1 ratio to receive either test product A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Mode of Usage: Twice a day on clean skin Route of Administration: Topical application.
  Interventions: Other: Placebo
- Anti-Ageing and Skin Brightening Gel (Experimental): Mode of Usage: Twice a day on clean skin Route of Administration: Topical application.
  Interventions: Other: Anti-Ageing and Skin Brightening Gel

INTERVENTIONS:
Other: Placebo — Placebo Comparator
  Arms: Placebo
Other: Anti-Ageing and Skin Brightening Gel — Anti-Ageing and Skin Brightening Gel.
  Arms: Anti-Ageing and Skin Brightening Gel

SUMMARY:
This is a Randomized, Interventional, Prospective, Double Blind, Two Arm, Comparative, Parallel, Placebo-Controlled, Safety and Efficacy Study of Anti-Ageing and Skin Brightening Gel.

Total of 44 adult female subjects (22 Subjects/Arm) of age 35 - 55 years will be enrolled to get 40 completed subjects (20 Subjects/Arm)

DETAILED DESCRIPTION:
There will be a total of 3 visits in the study. The subject will be instructed to visit the facility as per the below visits Visit 01 (Day 01): Screening, Enrolment and Treatment Start Phase (Week 00) Visit 02 (Day 30): Treatment Phase (Week 04) Visit 03 (Day 60): End of Study (Week 08) The potential subjects will be screened as per the inclusion and exclusion criteria only after obtaining written informed consent. Subjects will be asked to not wear any makeup on the face on screening day.

Assessment of efficacy parameters before test products usage will be done on Day 01 after enrolment and after test products usage will be done on Day 30 (± 2 days) and Day 60 (± 2 days) as listed-below.

* PGA scoring using Griffiths scale - skin dryness, redness, fine wrinkling/lines, coarse wrinkling/lines, laxity, roughness and sallowness.
* Glogau skin age.
* Skin pigmentation scoring.
* Skin elasticity: Cutometer Dual MPA 580.
* Skin colorimeter CL 400: CIE L*, a* b*, ITA angle, skin brightness, skin pigmentation reduction.
* Skin Glossymeter GL200 - skin glow.
* Visioscan (C+K instrument): crow's feet area wrinkles, fine lines, skin texture - roughness, dryness, wrinkles, smoothness.
* Digital photographs: facial photographs before test products usage on day 1 and post-usage at day 60.
* Image-pro software - image analysis day 01 vs day 60 - wrinkles, fine lines, pores.
* Subjective product perception assessment regarding the test product's effect on skin firmness, appearance, radiance, acne or skin breakouts, glowing skin tone, blemishes and dark skin patches removal etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 35 to 55 years (both inclusive) at the time of consent.
2. Sex: Healthy and non-pregnant/non-lactating females.
3. Subjects who are generally in good health as determined by/form recent medical history.
4. Female of child bearing capacity must have a self-reported negative pregnancy test.
5. Subjects having mild to moderate crows' feet wrinkles.
6. Subjects having a score of at least "mild skin aging" based on PGA at screening visit.
7. Subjects having a score of at least "mild skin pigmentation" based on Skin Pigmentation Score at screening visit.
8. Subjects having Glogau Skin Age II or III as assessed by the Dermatologist/ Dermatologist Trained Evaluator.
9. Subjects who are willing to forgo cosmetic procedures for the duration of the study.
10. Subjects who are able to follow their normal skin care routines and to refrain from introducing any new skin care products during the study.
11. Subjects who are willing not to introduce any new soaps, cleansers, lotions, creams, or any other face products etc. for the duration of the study.
12. Subjects who are willing to give written informed consent and are willing to follow the study procedure.
13. Subjects who commit not to use medicated/ prescription anti-ageing and skin brightening products or any other anti-ageing and skin brightening products other than the test products for the entire duration of the study.
14. Subjects who are willing to use test products throughout the study period.

Exclusion Criteria:

1. Subjects having a history of allergy or sensitivity to the test treatments ingredients.
2. Subjects who have pre-existing or dormant dermatologic conditions (e.g., psoriasis rashes, eczema, seborrheic dermatitis, acne or any other) that could interfere with the outcome of the study as determined by the Investigator.
3. Subjects who have used any systemic therapy with chronic antibiotic therapy, retinoids, and/or oral steroids during the 4 weeks prior to the start or anticipates having to use at any point during the study.
4. Subjects who have applied any topical retinoids within 2 weeks of the screening visit or anticipates having to use at any point during the study.
5. Subjects not willing to avoid unprotected sun or other UV radiation exposure during the study period.
6. Subjects having a history of alcohol or drug addiction.
7. Subjects who have used any systemic therapy with chronic antibiotic therapy, retinoids, and/or oral steroids during the 4 weeks prior to the start or anticipates having to use at any point during the study.
8. Subjects who have applied any topical retinoids or glutathione within 2 weeks of the screening visit or anticipates having to use at any point during the study.
9. Subjects not willing to avoid unprotected sun or other UV radiation exposure during the study period.
10. Subjects who are currently pregnant/breastfeeding or planning to become pregnant during the study period.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Skin Elasticity | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in Skin Elasticity from "before test product usage" and "after test product usage" using Cutometer Dual MPA 580
Change in CIE L*, a* b*, ITA (Individual Topography Angle), skin brightness, skin pigmentation | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in CIE L*, ITA angle, a* and b* from "before test product usage" and "after test product usage" using Skin Colorimeter CL 400.
Change in Skin Glow | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in Skin Glow from "before test product usage" and "after test product usage" using Skin Glossymeter GL 200.
Change in crow's feet area wrinkles, fine lines | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in crow's feet area wrinkle, fine line from "before test product usage" and "after test product usage" using Visioscan VC 20
Change in Skin texture (wrinkles, fine lines, roughness, dryness, wrinkles, and smoothness) of skin | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in Skin texture (wrinkles, fine lines, roughness, dryness, wrinkles, and smoothness) of skin from "before test product usage" and "after test product usage" using Visioscan VC 20
Change in facial photographs | From baseline (Day 01) before usage of test products to Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in facial photographs from "before test product usage" and "after test product usage" using digital photographs.
Change in wrinkles, fine lines and pores | From baseline (Day 01) before usage of test products to Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in wrinkles, fine lines and pores from "before test product usage" and "after test product usage" using Image-pro Software.

SECONDARY OUTCOMES:
Change in Physician Global Assessment (PGA) Score | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of test treatment in terms of change in PGA scores i.e. dryness, redness, fine lines, coarse wrinkle, laxity, roughness, and sallowness by using Griffith scale Where 0= No appearance and 9= Severe
Change in Level of skin photodamage | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in level of photodamage using Glogau skin age
Change in skin pigmentation | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the effectiveness of the test products in terms of change in skin pigmentation using skin pigmentation scoring. Scoring Scale:(0-absent, 1-mild, 2-moderate, 3-severe)
Assessment of Consumer Perception | From baseline (Day 01) before usage of test products to Day 30 (±2 days) and Day 60 (±2 days) post-usage of test products
  To assess the consumer perception of the test products regarding the test product's effect on skin firmness, appearance, radiance, acne or skin breakouts, glowing skin tone, blemishes and dark skin patches removal using questionnaire. Scoring Scale: (1- strongly disagree, 2-disagree, 3-neither agree nor disagree, 4-agree, 5-strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, Principal Investigator — NovoBliss Research Private Limited
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No